CLINICAL TRIAL: NCT01613326
Title: A 12-week Treatment, Randomized, Blinded, Double-dummy, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of NVA237 (50 µg o.d.) Compared to Tiotropium (18 µg o.d.) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy, Safety, and Tolerability of NVA237 Compared to Tiotropium in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: GLOW5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2314; 2011-000960-93 (EudraCT Number)
Record Dates: First submitted 2012-02-17; First posted 2012-06-07 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 (Experimental): NVA237 50 μg once a day and placebo to tiotropium once a day during 85 days. Salbutamol/albuterol was provided as rescue medication.
  Interventions: Drug: NVA237; Drug: Placebo to tiotropium; Drug: salbutamol/albuterol
- Tiotropium (Active Comparator): Tiotropium 18 μg once a day and placebo to NVA237 once a day during 85 days. Salbutamol/albuterol was provided as rescue medication.
  Interventions: Drug: Tiotropium; Drug: Placebo to NVA237

INTERVENTIONS:
Drug: NVA237 — NVA237 50 μg inhalation capsules once a day, delivered via SDDPI
  Arms: NVA237
Drug: Tiotropium — Tiotropium 18 μg once a day delivered via HandiHaler® device
  Arms: Tiotropium
Drug: Placebo to tiotropium — Placebo to tiotropium 18 μg o.d. once a day delivered via HandiHaler® device.
  Arms: NVA237
Drug: Placebo to NVA237 — Placebo to NVA237 50 μg once a day delivered via SDDPI
  Arms: Tiotropium
Drug: salbutamol/albuterol — salbutamol/albuterol given as a rescue medication via inhaler when needed
  Arms: NVA237

SUMMARY:
This study compared the efficacy and safety of NVA237 with tiotropium in patients with moderate to severe COPD. Tiotropium belongs to the same drug class as NVA237.

DETAILED DESCRIPTION:
This was a randomized, blinded, double-dummy, parallel-group 12-week study to assess the efficacy, safety, and tolerability of NVA237 (50 μg o.d.) compared to tiotropium (18 μg o.d.) in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable COPD (Stage II or Stage III) according to the current GOLD Guidelines (GOLD 2010).
* Patients with a post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) ≥ 30% and < 80% of the predicted normal, and a post-bronchodilator FEV1/ Forced Vital Capacity (FVC) < 0.70 at screening
* Current or ex-smokers who have a smoking history of at least 10 pack years (e.g. 10 pack years = 1 pack/day x 10 yrs, or ½ pack/day x 20 yrs).
* Symptomatic patients, according to daily electronic diary data between Visit 2 (Day -14) and Visit 3 (Day 1), with a total score of 1 or more on at least 4 of the last 7 days prior to Visit 3.

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Patients who, in the judgment of the investigator, or the responsible Novartis personnel, have a clinically relevant laboratory abnormality or a clinically significant condition before Visit 1.
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment or urinary retention. (BPH patients who are stable on treatment can be considered).
* Patients receiving medications in the classes listed in the protocol as prohibited.

Other protocol-defined inclusion/exclusion criteria apply and can be found in the study protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (63):
- Canada (4):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
- Croatia (3):
  - Novartis Investigative Site, Sisak, Croatia
  - Novartis Investigative Site, Zagreb, Croatia
  - Novartis Investigative Site, Zagreb
- Czechia (6):
  - Novartis Investigative Site, Cvikov, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Rudná, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Žatec, Czech Republic
- Estonia (3):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Paide
  - Novartis Investigative Site, Tallinn
- France (4):
  - Novartis Investigative Site, Beuvry, France
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Reims
- Germany (9):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- India (6):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Chennai - Tamil Nadu, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Utena
  - Novartis Investigative Site, Vilnius
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Bulacan, Philippines
  - Novartis Investigative Site, Manila, Philippines
  - Novartis Investigative Site, Quezon City
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- South Africa (2):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Gatesville
- South Korea (5):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Taiwan (5):
  - Novartis Investigative Site, Chiayi City, Taiwan
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei County, Taiwan
  - Novartis Investigative Site, Chiayi City

REFERENCES:
- [Derived] Chapman KR, Beeh KM, Beier J, Bateman ED, D'Urzo A, Nutbrown R, Henley M, Chen H, Overend T, D'Andrea P. A blinded evaluation of the efficacy and safety of glycopyrronium, a once-daily long-acting muscarinic antagonist, versus tiotropium, in patients with COPD: the GLOW5 study. BMC Pulm Med. 2014 Jan 17;14:4. doi: 10.1186/1471-2466-14-4. PMID 24438744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 980 patients were screened, and 657 were randomized (327 to NVA237 and 330 to tiotropium).
Pre-assignment Details: Patients meeting the eligibility criteria were randomized to receive NVA237 50 μg o.d. or tiotropium 18 μg o.d. in a 1:1 ratio. Patients were stratified according to their smoking status (current / ex-smoker).
Period: Overall Study
Arm/Group | NVA237 | Tiotropium
Started | 327 | 330
Completed | 314 | 316
Not Completed | 13 | 14
Not completed — Adverse Event | 7 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Abnormal test procedure result(s) | 2 | 0
Not completed — inability to use device | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | Tiotropium | Total
Number analyzed (Participants) | 327 | 330 | 657
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (7.98) | 63.7 (8.02) | 63.5 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 82 | 172
  Male | 237 | 248 | 485

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 12 Weeks of Treatment (Non-inferiority Analysis)
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 was defined as the mean of two measurements at 23hours 15min and 23 hours 45min post dosing. ANCOVA model: Trough FEV1 = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center (region). This analysis excluded values within 6 hours of rescue medication use or 7 days of systemic corticosteroid use.
Time Frame: Week 12
Population: The per-protocol set included all randomized patients who received at least one dose of study drug, with available data and without any major protocol deviations or who did not take study drug as per protocol in the 14 day period prior to trough.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 295 | 289
Liters | 1.405 (0.0173) | 1.405 (0.0170)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 12 Weeks of Treatment (Analysis of Superiority)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 was defined as the mean of two measurements at 23h 15min and 23h 45min post dosing. ANCOVA model: Trough FEV1 = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). This analysis excluded values within 6 hours of rescue medication use or 7 days of systemic corticosteroid.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 316 | 319
Liters | 1.398 (0.0154) | 1.393 (0.0149)

3. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score After 4 Weeks and 12 Weeks of Treatment
Description: Transition Dyspnea Index (TDI) captures changes from baseline. The TDI score is based on three domains with each domain scored from -3 (major deterioration) to +3 (major improvement), to give an overall score of -9 to +9, a negative score indicating a deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline.
  ANCOVA model: TDI focal score = treatment + Baseline dyspnea index (BDI) + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: Weeks 4 and 12
Population: The per-protocol set included all randomized patients who received at least one dose of study drug, with available data and without any major protocol deviations.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 290 | 287
Units on a scale
  Week 4 (n= 289, 287) | 2.209 (0.2957) | 2.086 (0.2945)
  Week 12 (n= 290, 285) | 1.990 (0.3169) | 2.178 (0.3159)

4. Secondary Outcome: St. George's Respiratory Questionnaire Total Score After 12 Weeks of Treatment
Description: St. George's Respiratory Questionnaire (SGRQ) is a health related quality of life questionnaire consisting of 51 items in three areas: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). The total score is 0 to 100 with a higher score indicating poorer health status. ANCOVA model: SGRQ total score = treatment + baseline SGRQ score + baseline ICS use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center (region).
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 290 | 285
Units on a scale | 39.42 (1.313) | 38.77 (1.306)

5. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication Used Over the 12 Week Treatment
Description: A day with no rescue medication use is defined from the diary data as any day where the patient recorded no rescue medicine use during the previous 12 hours.
  Baseline mean daily, daytime and nighttime (combined) number of puffs is defined as the average of the respective number of puffs. Only patients with a value at both baseline and post-baseline visits were included.
Time Frame: Baseline and Day 1 to Week 12
Population: The per-protocol set included all randomized patients who received at least one dose of study drug, with a value at both baseline and post-baseline visits were included.
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 296 | 290
puffs
  Baseline | 4.09 (3.816) | 4.10 (3.791)
  Day 1 to week 12 | 2.76 (2.768) | 2.84 (2.934)

6. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 1 and Week 4
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
  Trough FEV1 is defined as the average of the post-dose 23 h 15 min and the 23 h 45 min FEV1 values. Trough assessments taken outside 22 h 45 min - 24 h 15 min are excluded from this analysis.
  ANCOVA model: Trough FEV1 = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: Day 1 and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 296 | 288
Liters
  Day 1 (n=296, 288) | 1.385 (0.0124) | 1.386 (0.0122)
  Week 4 (n=284, 280) | 1.416 (0.0163) | 1.416 (0.0160)

7. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) During 5 Min to 4 Hours Post-dose, at Day 1 and Week 12
Description: Spirometry was conducted according to internationally accepted standards. Peak FEV1 is the maximum FEV1 recorded during first 4 hours post dose. ANCOVA model: Peak FEV1 = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center (region). Center is included as a random effect nested within region. This analysis excludes values within 6 hours of rescue medication use or 7 days of systemic corticosteroid use.
Time Frame: 5 min to 4 hours post-dose at Day 1 and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 298 | 292
Liters
  Day 1 (n= 298, 292) | 1.575 (0.0123) | 1.520 (0.0121)
  Week 12 (n= 290, 282) | 1.577 (0.0166) | 1.553 (0.0163)

8. Secondary Outcome: Inspiratory Capacity (IC) at Each Time-point, by Visit
Description: IC was measured with spirometry conducted according to internationally accepted standards. ANCOVA model: IC = treatment + baseline IC + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: (25 min, 1 h 55 min, 3 h 55 min, 23 h 40 min Day 1), (-20 min, 25 min, 23 h 40 min Week 4),(-20 min, 25 min, 1 h 55 min, 3 h 55 min, 23 h 40 min Week 12)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 216 | 214
Liters
  Day 1, 25 min (n= 216, 214) | 2.378 (0.0263) | 2.300 (0.0253)
  Day 1, 1 h 55 min (n= 212, 208) | 2.433 (0.0313) | 2.335 (0.0298)
  Day 1, 3 h 55 min (n= 211, 207) | 2.343 (0.0325) | 2.309 (0.0317)
  Day 1, 23 h 40 min (n= 213, 212) | 2.247 (0.0306) | 2.244 (0.0294)
  Week 4, -20 min (n= 204, 204) | 2.231 (0.0342) | 2.240 (0.0326)
  Week 4, 25 min (n= 201, 200) | 2.335 (0.0330) | 2.334 (0.0312)
  Week 4, 23 h 40 min (n=199,205) | 2.284 (0.0362) | 2.289 (0.0347)
  Week 12, -20 min (n= 205, 204) | 2.198 (0.0408) | 2.227 (0.0394)
  Week 12, 25 min (n= 215, 205) | 2.292 (0.0397) | 2.280 (0.0385)
  Week 12, 1 h 55 min (n= 213, 203) | 2.344 (0.0432) | 2.289 (0.0421)
  Week 12, 3 h 55 min (n= 203, 207) | 2.313 (0.0395) | 2.275 (0.0374)
  Week 12, 23 h 40 min (n= 208, 206) | 2.228 (0.0390) | 2.262 (0.0373)

9. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at Each Time-point by Visit
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 was analyzed using Analysis of Covariance (ANCOVA) model: FEV1 = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: (5,15,30 min, 1, 2,3,4 h, 23h 15 min and 23h 45 min postdose of Day 1), (-45, -15 min predose, 5,15,30 min, 1h, 23h 15 min and 23h 45 min postdose of Week 4), (-45, -15 min predose, 5,15,30 min, 1, 2, 3,4 h, 23h 15 min and 23h 45 min postdose of Week 12)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 291 | 286
Liters
  Day 1, 5 min (n= 283, 278) | 1.382 (0.0087) | 1.331 (0.0086)
  Day 1, 15 min (n= 282, 276) | 1.428 (0.0086) | 1.365 (0.0084)
  Day 1, 30 min (n= 285, 281) | 1.442 (0.0104) | 1.379 (0.0102)
  Day 1, 1 hour (n= 291, 286) | 1.482 (0.0111) | 1.419 (0.0109)
  Day 1, 2 hours (n= 290, 286) | 1.517 (0.0127) | 1.454 (0.0126)
  Day 1, 3 hours (n= 291, 285) | 1.527 (0.0141) | 1.471 (0.0138)
  Day 1, 4 hours (n= 285, 281) | 1.490 (0.0137) | 1.448 (0.0135)
  Day 1, 23 h 15 min (n= 289, 279) | 1.384 (0.0127) | 1.384 (0.0124)
  Day 1, 23 h 45 min (n= 285, 278) | 1.381 (0.0139) | 1.379 (0.0140)
  Week 4, -45 min (n= 280, 280) | 1.403 (0.0145) | 1.391 (0.0140)
  Week 4, -15 min (n= 278, 279) | 1.388 (0.0146) | 1.393 (0.0139)
  Week 4, 5 min (n= 277, 274) | 1.422 (0.0165) | 1.423 (0.0160)
  Week 4, 15 min (n= 271, 270) | 1.459 (0.0163) | 1.466 (0.0159)
  Week 4, 30 min (n= 272, 276) | 1.454 (0.0179) | 1.442 (0.0175)
  Week 4, 1 hr (n= 280, 282) | 1.513 (0.0152) | 1.494 (0.0147)
  Week 4, 23 h 15 min (n= 278, 276) | 1.422 (0.0171) | 1.417 (0.0167)
  Week 4, 23 h 45 min (n= 274, 276) | 1.418 (0.0165) | 1.416 (0.0162)
  Week 12, -45 min (n= 286, 279) | 1.394 (0.0176) | 1.380 (0.0174)
  Week 12, -15 min (n= 283, 279) | 1.377 (0.0168) | 1.370 (0.0165)
  Week 12, 5 min (n= 283, 271) | 1.430 (0.0182) | 1.411 (0.0181)
  Week 12, 15 min (n= 275, 271) | 1.440 (0.0168) | 1.423 (0.0163)
  Week 12, 30 min (n= 282, 278) | 1.461 (0.0168) | 1.432 (0.0163)
  Week 12, 1 hr (n= 286, 279) | 1.500 (0.0164) | 1.475 (0.0160)
  Week 12, 2 hours (n= 278, 277) | 1.507 (0.0173) | 1.484 (0.0169)
  Week 12, 3 hours (n= 281, 279) | 1.506 (0.0179) | 1.484 (0.0175)
  Week 12, 4 hours (n= 282, 280) | 1.473 (0.0187) | 1.462 (0.0183)
  Week 12, 23 h 15 min (n= 276, 266) | 1.414 (0.0185) | 1.422 (0.0183)
  Week 12, 23 h 45 min (n= 278, 276) | 1.415 (0.0183) | 1.420 (0.0180)

10. Secondary Outcome: Forced Vital Capacity (FVC) at Each Time-point by Visit
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. ANCOVA model: FVC = treatment + baseline FVC + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 291 | 286
Liters
  Day 1, 5 min (n= 283, 278) | 2.925 (0.0249) | 2.874 (0.0247)
  Day 1, 15 min (n= 282, 276) | 3.004 (0.0281) | 2.954 (0.0280)
  Day 1, 30 min (n= 285, 281) | 3.036 (0.0277) | 2.991 (0.0274)
  Day 1, 1 hour (n= 291, 286) | 3.036 (0.0298) | 3.006 (0.0296)
  Day 1, 2 hours (n= 290, 286) | 3.061 (0.0314) | 3.029 (0.0312)
  Day 1, 3 hours (n= 291, 285) | 3.135 (0.0334) | 3.111 (0.0329)
  Day 1, 4 hours (n= 285, 281) | 3.073 (0.0305) | 3.046 (0.0301)
  Day 1, 23 h 15 min (n= 289, 279) | 2.911 (0.0287) | 2.951 (0.0284)
  Day 1, 23 h 45 min (n= 285, 278) | 2.942 (0.0279) | 2.951 (0.0279)
  Week 4, -45 min (n= 280, 280) | 2.933 (0.0338) | 2.943 (0.0331)
  Week 4, -15 min (n= 278, 279) | 2.879 (0.0356) | 2.898 (0.0345)
  Week 4, 5 min (n= 277, 274) | 2.954 (0.0363) | 2.997 (0.0354)
  Week 4, 15 min (n= 271, 270) | 3.021 (0.0378) | 3.058 (0.0372)
  Week 4, 30 min (n= 272, 276) | 3.005 (0.0413) | 3.011 (0.0407)
  Week 4, 1 hr (n= 280, 282) | 3.068 (0.0381) | 3.093 (0.0374)
  Week 4, 23 h 15 min (n= 278, 276) | 2.982 (0.0364) | 3.013 (0.0359)
  Week 4, 23 h 45 min (n= 274, 276) | 2.953 (0.0372) | 2.978 (0.0366)
  Week 12, -45 min (n= 286, 279) | 2.889 (0.0416) | 2.905 (0.0415)
  Week 12, -15 min (n= 283, 279) | 2.827 (0.0358) | 2.837 (0.0355)
  Week 12, 5 min (n= 283, 271) | 2.929 (0.0403) | 2.953 (0.0403)
  Week 12, 15 min (n= 275, 271) | 2.945 (0.0370) | 2.963 (0.0364)
  Week 12, 30 min (n= 282, 278) | 2.963 (0.0374) | 2.982 (0.0367)
  Week 12, 1 hr (n= 286, 279) | 3.011 (0.0377) | 3.009 (0.0373)
  Week 12, 2 hours (n= 278, 277) | 3.008 (0.0390) | 3.012 (0.0386)
  Week 12, 3 hours (n= 281, 279) | 3.014 (0.0404) | 3.018 (0.0399)
  Week 12, 4 hours (n= 282, 280) | 2.964 (0.0404) | 2.977 (0.0398)
  Week 12, 23 h 15 min (n= 276, 266) | 2.923 (0.0403) | 2.953 (0.0404)
  Week 12, 23 h 45 min (n= 278, 276) | 2.929 (0.0436) | 2.955 (0.0434)

11. Secondary Outcome: Standardized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) (5 Min-4 h) Post-dose
Description: Forced Expiratory Volume in one second (FEV1) was measured with spirometry conducted according to internationally accepted standards.
  Area Under the Curve (AUC) is calculated using the trapezoidal rule using the existing FEV1 measurements (i.e., the missing FEV1 measurements are not interpolated).
  ANCOVA model: FEV1 AUC = treatment + baseline FEV1 + baseline Inhaled corticosteroid (ICS) use (Yes/No) + FEV1 reversibility components + baseline smoking status + region + center(region). Center is included as a random effect nested within region.
Time Frame: Day 1 and week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 298 | 292
Liters
  Day 1 (n=298, 292) | 1.496 (0.0109) | 1.438 (0.0107)
  Week 12 (290, 282) | 1.493 (0.0164) | 1.470 (0.0160)

12. Secondary Outcome: Event Free Rate at Weeks 4, 8 and 12 After Treatment
Description: Event free rate was calculated as a percentage of participants who did not experience any moderate or severe COPD exacerbation leading to hospitalization/treatment with systemic corticosteroids/treatment with antibiotics. The event free rate reflects the percent of patients who did NOT have an exacerbation by 4, 8 and 12 weeks. Event-free rates are calculated at the end of the specified weeks (i.e. Day 29, Day 57 and Day 85) by the Kaplan Meier method.
Time Frame: Weeks 4, 8 and 12
Population: The per-protocol set included all randomized patients who received at least one dose of study drug, with available data and without any major protocol deviations and described as patients with moderate to severe exacerbations were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 29 | 22
percentage of participants
  Week 4 | 95.6 [92.6 to 97.4] | 96.6 [93.7 to 98.1]
  Week 8 | 92.9 [89.3 to 95.3] | 93.8 [90.4 to 96.1]
  Week 12 | 90.2 [86.1 to 93.2] | 92.4 [88.8 to 95.0]

13. Secondary Outcome: Mean Daily, Daytime and Nighttime (Combined) Symptom Scores Over the 12 Week Treatment Period
Description: Participants completed eDiaries providing scores 0 to 3 for symptoms: Cough and wheeze (none, mild, moderate, severe); sputum volume (none, less than 5 mL, 5-25 mL, >25 mL); sputum color (none, white-grey, yellow, green); lowest level of activity causing breathlessness (never or only when running, when walking uphill or upstairs, when walking on flat ground, at rest). Symptoms in the morning, for the previous night (no waking due to symptoms, woke up once due to symptoms, woke up more than once due to symptoms, woke up frequently or could not sleep due to symptoms). Symptoms experienced during the day that had prevented them for performing normal activities (not at all, a little, quite a lot, completely). The mean change from baseline in the total scores and in the individual scores was summarized by treatment. Only participants with a value at both baseline and post-baseline were included. Possible total scores 0-18 (night); 0-36 (day). A higher score means worsening of symptoms.
Time Frame: 12 weeks
Population: The per-protocol set included all randomized patients who received at least one dose of study drug. Only patients with a value at both baseline and post-baseline are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 296 | 290
units on a scale
  Baseline | 7.21 (2.539) | 6.90 (2.627)
  Day 1 to Week 12 | 5.96 (2.469) | 5.96 (2.531)

ADVERSE EVENTS:
Arm/Group | NVA237 | Tiotropium
Serious Adverse Events (participants affected / at risk) | 11/327 | 13/330
Other Adverse Events (participants affected / at risk) | 48/327 | 54/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=327) | Tiotropium (N=330)
Cardiac failure (Cardiac disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=327) | Tiotropium (N=330)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 48 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.